CLINICAL TRIAL: NCT02968862
Title: Preemptive Analgesia for Postoperative Pain Relief in Thoraco-lumbo-sacral Spine Surgery: a Double-blinded Randomized Controlled Trial
Brief Title: Comparing Analgesia for Postoperative Pain Relief in Spine Surgery
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Linda S Aglio, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2010P000602
Record Dates: First submitted 2016-11-10; First posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: observational — The study will involve adult patients undergoing elective thoracolumbar-sacral spine surgery involving 1-5 spine levels, at the Brigham and Women's hospital that have an anticipated post surgical hospital stay of one to three days. These patients will be randomly assigned by the BWH Investigational Drug Service to one of three different groups, each consisting of 33 patients. This is an observational studies with subjects in which biomedical and/or health outcomes are assessed in pre-defined groups of individuals. Subjects in the study may receive a therapeutic intervention, but the investigator does not assign specific interventions to the subjects of the study.

SUMMARY:
The study will involve adult patients undergoing elective thoracolumbar-sacral spine surgery involving 1-5 spine levels, at the Brigham and Women's hospital that have an anticipated post surgical hospital stay of one to three days. These patients will be randomly assigned by the BWH Investigational Drug Service to one of three different groups, each consisting of 33 patients:

• Group 1 will be patients that will receive epidural hydromorphone 0. 5mg and bupivicaine 6.25 mg for a total volume of 10 ml.

* Group 2 patients will receive hydromorphone 0.5 mg in preservative free saline for a total volume of 10ml.
* Group 3 patients will receive 10 ml of preservative free saline and this will serve as the control group.

DETAILED DESCRIPTION:
The study will involve adult patients undergoing elective thoracolumbar-sacral spine surgery involving 1-5 spine levels, at the Brigham and Women's hospital that have an anticipated post surgical hospital stay of one to three days. These patients will be randomly assigned by the BWH Investigational Drug Service to one of three different groups, each consisting of 33 patients:

• Group 1 will be patients that will receive epidural hydromorphone 0. 5mg and bupivicaine 6.25 mg for a total volume of 10 ml.

* Group 2 patients will receive hydromorphone 0.5 mg in preservative free saline for a total volume of 10ml.
* Group 3 patients will receive 10 ml of preservative free saline and this will serve as the control group.

Exclusion criteria would be:

1. Anyone unable to sign consent
2. Pregnant patients
3. Non-elective surgery
4. Allergy to any of the study drugs or equipment
5. Any medical condition not compatible with the use of epidural anesthesia such as multiple sclerosis
6. Any patient with a rash at the surgical site or for cerebrospinal leak repair
7. Any patient who is currently anticoagulated for any reason (drugs or pathologic condition)
8. Patient who in the opinion of the Investigator may not be a suitable candidate for this study All subjects will be provided information about the study at their surgical appointment.

The study coordinator will approach the patient with permission from the surgeon and introduce the study and one of the co- investigators will explain the study to the patient.

The investigator will subsequently review their eligibility and the inclusion criteria (thoracolumbar-sacral spine surgery, hospital stay greater than one to three days, and no history of allergy to local anesthetics or opioids) and the exclusion criteria (documented allergy, pregnant female, minor, or ongoing cerebrospinal fluid leak coagulation status). If the subject continues to meet all the criteria, the investigator will explain the study with the patient and answer all questions. Thereafter, the patients will be provided the consent forms for their review and a 24/7 contact number for any questions regarding this study.

All patient questions will be answered and informed consent will be obtained by the investigator at this time. The patient will be provided with contact information. A co-investigator will be available to answer questions a on a 24-hour basis. It will be explained to the patient that they will be permitted to withdraw from the study at any time for any reason until the day of their surgery.

On arrival at the preoperative area, the patient will be assigned a code by one of the investigators. The BWH Investigational Drug service will be utilized to ensure randomization and proper preparation and storage of the study drug and the safety of the subjects.

The subjects will be randomized to one of three groups. Subjects will be randomized by the BWH Investigational Drug Service. The surgeon will be informed of the patient's participation in the study but not the study group to which they are assigned.

Prior to premedication, all patients will be made familiar with the use of the 10-cm visual analog scale (VAS), with 0 = no pain, and 10 = worst pain imaginable. The baseline (VAS) score will be recorded.

All routine standard practices for surgery, anesthesia and perioperative care will be followed.

All patients will be premedicated with (0.025 - 0.05mg/kg) of midazolam. An epidural will be placed in the preoperative area by the anesthesiologist.

■ Patients will be randomized. Patients belonging to Group 1 will receive epidural hydromorphone 0.5mg and bupivicaine 6.25 mg for a total volume of 10 ml; Group 2 patients will receive hydromorphone 0.5 mg in preservative free saline for a total volume of 10ml. Group 3 will receive 10 ml of preservative free saline and this will be the control group.

The epidural will be placed by the anesthesiologist two vertebral levels above the level of surgery.

A standard total intravenous anesthesia (TIVA) protocol will be followed since somatosensory and motor evoked potentials are routinely monitored throughout the surgery in these cases.

Anesthesia will be induced with intravenous (IV) propofol (1.5-2.5mg/kg) and fentanyl (1.0-3.0 ug/kg). Tracheal intubation is facilitated with a neuromuscular blocking drug. The anesthetic will be maintained with a TIVA technique consisting of propofol and remifentanil infusions at 0.125 ug/kg/hr for maintenance, dilaudid 0.02-20.mg/kg begin titrating one hour after incision, with an oxygen/air mixture in 2:1 ratio. A BICS monitor will be used to monitor depth of anesthesia.

At the completion of the operation, the anesthesiologist will wake-up the patient and the patient will be transferred to the post anesthesia care unit (PACU).

The postoperative pain, sedation, nausea/vomiting, and constipation scores will be obtained and recorded by the Study Coordinator. This will be obtained by the visual analog scale (VAS) (enclosed) every 15 minutes up until 2 hours and on postoperative day one (24 hours). The type and time for the first demand for supplemental analgesia and the total amount will also be documented.

The primary endpoints of this study will be to determine the absolute reduction in pain scores among the groups.

Secondary endpoints would include the overall average pain control scores, the total amount of postoperative opioid consumption; the degree of opioid side effects for opioid consumption, the first demand for supplemental analgesia; the time to initial physical therapy participation, and the return to activities of daily living.

The patients will be assessed by questions that are part of the REDCAP database at their first post-operative visit about six weeks after their surgery. The questions will ask their general satisfaction with the study in relation to pain, nausea, vomiting and sedation using a 0-10 scale either during their post-op visit or by phone if they are not able to return to the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients
2. 8 years of age or older

Exclusion Criteria:

1. Anyone unable to sign consent
2. Pregnant patients
3. Non-elective surgery
4. Allergy to any of the study drugs or equipment
5. Any medical condition not compatible with the use of epidural anesthesia such as multiple sclerosis
6. Any patient with a rash at the surgical site or for cerebrospinal leak repair
7. Any patient who is currently anticoagulated for any reason (drugs or pathologic condition)
8. Patient who in the opinion of the Investigator may not be a suitable candidate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects will be provided information about the study at their surgical appointment.
  The study coordinator will approach the patient with permission from the surgeon and introduce the study and one of the co- investigators will explain the study to the patient.
  The investigator will review their eligibility and the inclusion criteria and the exclusion criteria. If the subject continues to meet all the criteria, the investigator will explain the study with the patient and answer all questions. Thereafter, the patients will be provided the consent forms for their review and a 24/7 contact number for any questions regarding this study.
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2009-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
low back pain | 24 hours
  The postoperative pain scores will be obtained and recorded by the Study Coordinator. This will be obtained by the visual analog scale (VAS) (enclosed) every 15 minutes up until 2 hours and on postoperative day one(24 hours). The type and time for the first demand for supplemental analgesia and the total amount will also be documented.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aglio LS, Abd-El-Barr MM, Orhurhu V, Kim GY, Zhou J, Gugino LD, Crossley LJ, Gosnell JL, Chi JH, Groff MW. Preemptive analgesia for postoperative pain relief in thoracolumbosacral spine operations: a double-blind, placebo-controlled randomized trial. J Neurosurg Spine. 2018 Dec 1;29(6):647-653. doi: 10.3171/2018.5.SPINE171380. Epub 2018 Sep 14. PMID 30215593